CLINICAL TRIAL: NCT02752178
Title: A Clinical Biomarker Study of Immunological Phenotypes Associated With Monoaminergic Anti-depressant Response, and the Brain and Cognitive Phenotypes Associated With Variation in Peripheral C-reactive Protein (CRP) Levels, in Patients With Major Depressive Disorder (MDD).
Brief Title: Peripheral Immunomarker Validation in Treatment-resistant Depression
Acronym: BIODEP
Status: Completed | Type: Observational
Sponsor: University of Cambridge (Other)
Collaborators: University of Oxford (Other); University of Glasgow (Other); University of Sussex (Other); King's College London (Other); Janssen, LP (Industry); H. Lundbeck A/S (Industry); GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Linda Pointon, Professor Edward T. Bullmore, University of Cambridge
Other Study IDs: 15/EE/0092
Record Dates: First submitted 2016-03-16; First posted 2016-04-26 (Estimated); Last update posted 2018-09-25 (Actual); Status verified 2018-09

CONDITIONS: Depressive Disorder, Major
Keywords: Depression; Major depressive disorder; MDD
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — 1-(2-(dodecyloxy)ethyl)pyrrolidine hydrochloride

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and saliva samples will be stored in a linked anonymised form for immunophenotyping and DNA analysis
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- DEP+MA+: Incompletely responsive patients (approximately N ~100) who are currently depressed after greater than 6 weeks of treatment with one or more monoaminergic antidepressants
  Interventions: Other: MA; Other: DEP
- DEP-MA+: Responsive patients (approximately N~50) who are not currently depressed after greater than 6 weeks of treatment with a monoaminergic antidepressant
  Interventions: Other: MA
- DEP+MA-: Untreated patients (approximately N~50) who are currently depressed but have not been treated with monoaminergic antidepressants in the previous 6 weeks
  Interventions: Other: DEP
- DEP-MA-: Healthy volunteers (approximately N~50) who have no personal history of depression requiring treatment with either monoaminergic antidepressants or other clinical interventions including psychotherapy

INTERVENTIONS:
Other: MA — Monoaminergic antidepressant use
  Groups: DEP+MA+; DEP-MA+
Other: DEP — Depression measured using the Hamilton Depression (HAM-D) questionnaire
  Groups: DEP+MA+; DEP+MA-

SUMMARY:
This is a study to characterise the role of inflammatory processes in depression. There is compelling evidence that inflammation is often associated with, and can cause, depression. It is currently less clear that antiinflammatory drugs have meaningful antidepressant effect. One of the goals is to identify the subset of depressed patients that is most likely to respond better to an antiinflammatory drug than to a conventional antidepressant. The investigators will therefore undertake a study of patients with a diagnosis of major depressive disorder including four groups: i) incompletely responsive patients who have demonstrated failure to respond consistently or completely to standard treatment, ii) those who have responded well to treatment and are not currently depressed, iii) untreated patients who are currently depressed, iv) healthy volunteers with no history of depression. Participants will undergo a clinical assessment, an interview with a trained member of the research team and will complete self-rated questionnaires. Investigators will collect blood and saliva samples to measure certain immune markers. They will also perform magnetic resonance imaging (MRI) scans to look for MRI markers in the brain and investigate brain inflammation in a subsample of these patients using positron emission topography (PET) and cerebrospinal fluid (CSF) sampling (also called lumbar puncture).

DETAILED DESCRIPTION:
The hypotheses are (i) that therapeutic resistance to monoaminergic (MA) antidepressant drugs is associated with peripheral biomarkers indicating abnormal activation of the innate immune system; and (ii) that peripheral inflammation, defined by blood levels of C-reactive protein (CRP), is associated with central nervous system inflammation and abnormal brain structure and function.

The objectives are to test these two hypotheses by collecting clinical, immunological and neuroimaging data on patients with depression (DEP+) recruited from a network of clinical research sites in the United Kingdom.

Primary objective:

To measure peripheral immunophenotypes in healthy volunteers (at least N=50) and 3 groups of depressed patients, categorised by their exposure and therapeutic response to monoaminergic antidepressants (up to N=200):

* Incompletely responsive patients (approximately N ~100) who are currently depressed after greater than 6 weeks of treatment with one or more monoaminergic antidepressants (DEP+MA+);
* Responsive patients (approximately N~50) who are not currently depressed after greater than 6 weeks of treatment with a monoaminergic antidepressant (DEP-MA+);
* Untreated patients (approximately N~50) who are currently depressed but have not been treated with monoaminergic antidepressants in the previous 6 weeks (DEP+MA-);
* Healthy volunteers (approximately N~50) who have no personal history of depression requiring treatment with either monoaminergic antidepressants or other clinical interventions including psychotherapy (DEP-MA-).

Secondary objective:

To measure brain and cognitive phenotypes in a subsample of up to N=100 depressed patients recruited, preferably from the primary cohort, on the basis of their CRP levels:

* Low CRP patients (N~45) will have CRP <= 3 mg/L
* High CRP patients (N~45) will have CRP > 3 mg/L
* Healthy volunteers (at least N=45).

All subjects in this sample will be assessed using structural and functional magnetic resonance imaging (MRI) and subjects providing additional specific consents will also be assessed using positron emission tomography (PET-MR), and/or lumbar puncture (LP) for cerebrospinal fluid (CSF) sampling.

ELIGIBILITY:
Inclusion Criteria:

* Major depressive disorder diagnosed by structured clinical interview in accordance with Diagnostic and Statistical Manual of Mental Disorders (DSM) criteria
* Aged 25-50 years inclusive
* HAM-D score at baseline

  1. DEP+MA+ subgroup > 13
  2. DEP+MA- subgroup > 17
  3. DEP-MA+ subgroup < 7
* Able and willing to give informed consent, including consent to sharing of clinical information with the participant's general practitioner
* Willing to abstain from strenuous exercise for 72 hours prior to assessment
* Able to write, speak and understand English

Exclusion Criteria:

* Life time history of bipolar disorder or nonaffective psychosis
* Concurrent medication likely to compromise the interpretation of immunological data (including, but not limited to corticosteroids, or any other substance to be determined by the Principal Investigator or delegate)
* Pregnancy or breast feeding
* Active alcohol or drug abuse or dependence in the last 6 months
* Participation in clinical trial of an investigational drug within the last 12 months
* Lifetime history of any serious medical disorder likely to compromise the interpretation of immunological data (including, but not limited to, immunological disorders, cardiovascular disorders, malignancies or infection, or any other condition to be determined by the Principal Investigator or delegate)

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: People with depression and healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 393 (Actual)
Dates: Start 2015-06; Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
C-reactive protein (CRP) levels (mg/l) | One year after last participant visit
Flow cytometric immunophenotype | One year after last participant visit
  The exact antibody panel will be developed during the research study

SECONDARY OUTCOMES:
Structural parameters of the brain | One year after last participant visit
  Measured using MRI. Specifically: larger grey matter volume loss, quantitative parameters (T1, T2), magnetization transfer, and the microstructure of grey and white matter
Response to stimulus | One year after last participant visit
  Specifically: functional MRI (fMRI) signatures obtained in an emotional face recognition and a reward processing task, respectively.
Microglial activation in the brain | One year after last participant visit
  Measured using Positron Emission Tomography (PET)
Pro-inflammatory (M1-like) phenotype-producing cytokines, such as interleukin (IL)-1, IL-6, and tumor necrosis factor (TNF)-α circulating in cerebrospinal fluid | One year after last participant visit

CONTACTS AND LOCATIONS:
Overall Officials: Edward T Bullmore, FRCPsych, Principal Investigator — University of Cambridge
Locations (5):
- United Kingdom (5):
  - University of Sussex, Brighton
  - University of Cambridge, Cambridge
  - University of Glasgow, Glasgow
  - King's College London, London
  - University of Oxford, Oxford

IPD SHARING:
Plan to Share IPD: Yes
All publications resulting from this study will be made available Open Access. Additionally, supporting research data will be also made available. This page will be updated with information about research outputs as soon as they become available.